CLINICAL TRIAL: NCT07211750
Title: Integrated Care for Older Adults With Major Depression and Physical Multimorbidity - The I-CONNECT
Acronym: I-CONNECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Goderis Geert, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: S70376
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-09

CONDITIONS: Multimorbidity; Older Adults (65 Years and Older); Mood Disorders; Depression - Major Depressive Disorder; Bipolar; Integrated Care
Keywords: Integrated care; Care coordination; Person-centered care; Shared decision-making; Self-management support; Multimorbidity; Depression; Bipolar disorder; Older adults; Quality of life
MeSH Terms: conditions — Mood Disorders; Depression; Bipolar Disorder | interventions — Multimorbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-CONNECT Integrated Care (Experimental): Participants receive the I-CONNECT care model: a trained care coordinator works with the participant, GP, psychiatrist, pharmacist, and specialists to create a personalized care plan, conduct a structured medication review, support shared decision-making and self-management, and provide regular follow-up (phone or in-person) to monitor progress and adjust care.
  Interventions: Other: integrated care intervention tailored to the needs of older adults leaving at home with mood disorders and multimorbidity in Leuven
- Standard Care (No Intervention): Participants continue their usual medical and mental healthcare. Their general practitioner and psychiatrist manage care as normally provided, without additional I-CONNECT coordination, medication review protocol, or structured follow-up from a care coordinator.

INTERVENTIONS:
Other: integrated care intervention tailored to the needs of older adults leaving at home with mood disorders and multimorbidity in Leuven — The six guiding principles are translated into practice through a structured six-step care model. Each step operationalizes one or more principles, ensuring that the model is consistently applied across patient trajectories. The program takes 12 months, with flexible contacts depending on patient's needs.
  Arms: I-CONNECT Integrated Care

SUMMARY:
The goal of this clinical trial is to learn if I-CONNECT (Integrated Care for Older Adults with Major Depression and Physical Multimorbidity) can improve the health and well-being of older adults with depression or bipolar disorder and at least two chronic physical conditions, such as diabetes or high blood pressure. It will also study if the care model improves how people experience their care, lowers treatment burden, and how well the program is delivered.

Researchers will compare two groups:

I-CONNECT group: participants receive care coordination, a personalized care plan, medication review, shared decision-making support, and regular follow-up from a care coordinator working with their GP, psychiatrist, pharmacist, and specialists.

Usual care group: participants continue with their normal healthcare from their GP and psychiatrist.

Participants will:

Receive either I-CONNECT or usual care, depending on their group

Complete questionnaires about their mood, quality of life, and care experience

Have their healthcare use (emergency visits and hospitalizations) tracked during the study

DETAILED DESCRIPTION:
Mood disorders, including depression and bipolar disorder, are common in older adults and frequently occur alongside multiple long-term physical health problems. This combination worsens quality of life, raises mortality risk, and increases healthcare use and costs. Despite the high burden, healthcare systems often provide fragmented care, with limited coordination between providers and underuse of mental health resources.

I-CONNECT is a person-centered integrated care model designed to address these challenges. It combines professional care coordination with structured medication review, active involvement of general practitioners, psychiatrists, pharmacists, and specialists, and support for self-management through shared decision-making. By bridging primary and mental healthcare, the model seeks to reduce fragmentation, strengthen continuity of care, and improve outcomes for older adults with complex needs.

Study Objectives The primary objective is to test whether I-CONNECT improves overall health outcomes compared with usual care. Secondary objectives are to examine participants' experiences of care, the burden of managing multiple health problems, and the impact on healthcare utilization.

Hypothesis

The investigators hypothesize that the I-CONNECT intervention will:

Improve both mental and physical health outcomes,

Reduce treatment burden and stress for participants,

Enhance satisfaction with care, and

Support a more efficient use of healthcare resources.

Implementation Evaluation In addition to effectiveness, the study will assess how I-CONNECT is implemented. Process measures will include fidelity to the care model, the amount of intervention delivered, and outcomes of medication reviews. Qualitative feedback from participants and providers will help identify barriers and facilitators to scale-up and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Clinical diagnosis of a mood disorder (depression or bipolar disorder)
* Currently receiving care from a psychiatrist
* At least two chronic physical health conditions
* Living independently at home in the Leuven region
* Ongoing care from both a general practitioner and a psychiatrist

Exclusion Criteria:

* Severe cognitive impairment (e.g., advanced dementia) that prevents participation in assessments or shared decision-making
* Inability to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Physical Component Summary (PCS) score from the SF-36 | Baseline and 6 months after randomization
  Change in the PCS score of the Short Form (SF-36) Health Survey, which reflects the physical health dimension of quality of life. A clinically meaningful improvement is defined as an increase of at least 5 points.
  Unit of Measure: Score (0-100)
Mental Component Summary (MCS) score from the SF-36 | Baseline and 6 months after randomization
  The MCS score from the Short Form-36 (SF-36) Health Survey will be used to evaluate the mental health dimension of quality of life. A clinically meaningful improvement is defined as an increase of at least 5 points.
  Unit of Measure: Score (0-100)

SECONDARY OUTCOMES:
Patient Assessment of Chronic Illness Care (PACIC) score | Baseline and 6 months after randomization
  Change in care experience measured by the Patient Assessment of Chronic Illness Care (PACIC). The PACIC contains 15 items across 5 domains. Each item is scored on a 5-point Likert scale (1 = "almost never" to 5 = "almost always"), and the total score is calculated as the mean of all item scores. Thus, the overall PACIC score ranges from 1 to 5, with higher scores indicating better alignment of care with the Chronic Care Model.
  Unit of Measure: Score (1-5)
Multimorbidity Treatment Burden Questionnaire (MTBQ) score | Baseline and 6 months after randomization
  Change in treatment burden measured by the Multimorbidity Treatment Burden Questionnaire (MTBQ). The MTBQ assesses the perceived difficulty of managing multiple health conditions and treatments, including medication, appointments, monitoring, and lifestyle changes. Scores range from 0 to 100, with higher scores indicating greater treatment burden.
Change in Physical Component Summary (PCS) score of the SF-36 over time | Baseline, 3 months, 6 months, and 12 months after randomization
  Description: Change in physical health-related quality of life measured by the PCS score of the SF-36 at multiple time points.
  Unit of Measure: Score (range: 0-100)
Change in Mental Component Summary (MCS) score of the SF-36 over time | Baseline, 3 months, 6 months, and 12 months
  Change in mental health-related quality of life measured by the MCS score of the SF-36 at multiple time points.
  Unit of Measure: Score (range: 0-100)
PACIC scores over time | Baseline, 3 months, 6 months, and 12 months after randomization
  Change in patient-reported care experience using the PACIC questionnaire at multiple time points to assess sustainability of effects.
MTBQ score over time | Baseline, 3 months, 6 months, and 12 months after randomization
  Change in treatment burden measured by the MTBQ at multiple time points to assess sustainability of effects.
Number of emergency room visits | 6 months and 12 months after randomization
  Description: Number of emergency room visits during the study period, based on patient report and confirmed by medical records when available.
  Unit of Measure: Count (visits per participant)
Number of hospital admissions | 6 months and 12 months after randomization
  Description: Number of hospital admissions during the study period, based on patient report and confirmed by medical records when available.
  Unit of Measure: Count (admissions per participant)

OTHER OUTCOMES:
Fidelity of intervention delivery | At study completion, 12 months following the randomization of the final enrolled patient.
  Adherence to delivering core components of the intervention, such as first appointment, life goal assessment, medication review, and proactive follow-up. Measured as the percentage of participants receiving each planned component. Electronic health records (EHRs) will also be reviewed to confirm delivery.
  Unit of Measure: Percentage of participants
Intervention dose | At study completion, 12 months after last patient randomized
  Intensity of the intervention received by patients, measured as the frequency of follow-up contacts compared with the planned individualized care schedule. Data obtained from EHRs.
  Unit of Measure: number of follow-up contacts per participant
Medication review outcomes: Number of new prescriptions | At study completion (12 months after last patient randomized)
  Number of new medications prescribed during the study period, based on EHR data.
  Unit of Measure: Count (prescriptions per participant)
Medication Review outcomes: Number of new deprescriptions | At study completion,12 months after last patient randomized
  Description: Number of medications deprescribed during the study period, based on EHR data.
  Unit of Measure: Count (prescriptions per participant)
Number of participants reporting medication side effects | Time Frame: At study completion,12 months after last patient randomized
  Description: Participants who experienced medication-related side effects during the study period, as reported in the EHR.
  Unit of Measure: Number of participants

CONTACTS AND LOCATIONS:
Locations (1):
- KU/UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided